CLINICAL TRIAL: NCT05100160
Title: Gabapentin for the Reduction of Opiate Use Following Pulmonary Resection (GROUP Trial)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: 0 patient accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-0653; NCI-2021-10727 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-09-22; First posted 2021-10-29 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Thoracic; Pulmonary Disease
MeSH Terms: conditions — Lung Diseases | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Experimental): used as part of a multimodal pain regimen (combination of drugs used to control pain
  Interventions: Drug: Gabapentin
- Placebo (Experimental): designed to be compared with a study drug to learn if the study drug has any real effect
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gabapentin — Given by PO
  Arms: Gabapentin
Other: Placebo — Given by PO
  Arms: Placebo

SUMMARY:
The aim of this study is to determine if the reduction in narcotic requirement following pulmonary resection with gabapentin is clinically significant when compared to the effect seen with placebo. We have defined clinically meaningful as a reduction by 30 Morphine equivalent doses (MED)

DETAILED DESCRIPTION:
Study Objectives:

The aim of this study is to determine if the reduction in narcotic requirement following pulmonary resection with gabapentin is clinically significant when compared to the effect seen with placebo. We have defined clinically meaningful as a reduction by 25% Morphine equivalent doses (MED) Secondary objectives are to evaluate the utility of gabapentin in reducing postoperative pain, reducing hospital length of stay, promoting faster return to baseline function (to be assessed by MDASI), preventing post thoracotomy pain syndrome (to be assessed by BPI), and reducing the rate of chronic opiate use among patients undergoing thoracic procedures.

1. Primary Endpoint

   The primary outcome will be the sum of the daily average morphine equivalent dose of opioids recorded from day of surgery (day 0) through 7 days after surgery, for a total of 8 days.
2. Secondary Endpoints

   * Time to resuming normal activities
   * Presence/absence of chronic pain at 3 and 6 months, measured by BPI
   * 30, 90, 180 day opiate use (Y/N)
   * MDASI on post-operative days 7, 30, 90, 180
   * Basic Pain Inventory (BPI) on post-operative days 1,2, 7, 30, 90, 180
   * Daily pain score during hospitalization
   * Length of hospital stay
   * Need for opioids at discharge
   * Whether medication is stopped prior to day 25, and if so when and for what reason.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Undergoing pulmonary resection (includes metastasectomy as well as anatomic resections)
* Must have device with email capabilities for follow up survey

Exclusion Criteria:

* Requiring narcotic pain medication or Gabapentin at the time of preoperative appointment or within 30 days of surgery
* Renal impairment requiring dialysis
* Allergy to Gabapentin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
The change in narcotic requirement following pulmonary resection with gabapentin is clinically significant when compared to the effect seen with placebo | through study completion, up to 8 days
  The sum of the daily average morphine equivalent dose of opioids recorded from day of surgery (day 0) through 7 days after surgery, for a total of 8 days

CONTACTS AND LOCATIONS:
Overall Officials: David Rice, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org